CLINICAL TRIAL: NCT02283918
Title: Study to Establish Patient-Matched Population Norms for the MS-COG
Brief Title: Observational Study to Establish Patient-Matched Population Norms for the Multiple Sclerosis Cognition Assessment Battery
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 999MS005
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Participants with education less than bachelor's degree: Participants are further divided into three sub-groups based on their age group Group 1: Participants aged between 25 to 34 years Group 2: Participants aged between 35 to 44 years Group 3: Participants aged between 45 to 58 years
- Participants with bachelor's degree or equivalent: Participants are further divided into three sub-groups based on their age group Group 1: Participants aged between 25 to 34 years Group 2: Participants aged between 35 to 44 years Group 3: Participants aged between 45 to 58 years

SUMMARY:
The primary objective of the study is to develop MS patient-matched healthy population norms for the Multiple Sclerosis Cognition Assessment Battery (MS-COG) that are representative of the United States (US), France, and Italy.

ELIGIBILITY:
Key Inclusion Criteria

1. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use confidential health information in accordance with national and local subject privacy regulations.
2. Must be in good health as determined by the Investigator, based on medical history, physical examination, and Screening evaluations.
3. Must be a native language speaker of the country where the study is being conducted.

Key Exclusion Criteria:

1. Neurological illnesses/conditions, such as motor or vocal tics (including a diagnosis of Tourette's syndrome), head trauma with significant loss of consciousness (>30 min), cerebral ischemia, carotid artery disease, epilepsy, brain tumor, dementia (including mild cognitive impairment and Alzheimer's disease), chronic meningitis, multiple sclerosis, pernicious anemia, normal-pressure hydrocephalus, HIV infection, Parkinson's disease, and Huntington's disease.
2. Medical illnesses/conditions that may affect brain function, such as untreated hypertension (blood pressure >140/100 mm Hg), cardiac disease, insulin-dependent diabetes mellitus, endocrine disorders, renal disease, glaucoma, and chronic obstructive pulmonary disease.
3. Major psychiatric disturbance according to the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (US) Axis I criteria [American Psychiatric Association 2013] and the International Statistical Classification of Diseases and Related Health Problems, 10th revision Axis I criteria (Europe) [WHO 2010].
4. History of developmental disorders.

Note: Other protocol defined Inclusion/ Exclusion criteria may apply.

Ages: 25 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This is a multinational, multicenter study that will be conducted in healthy adult volunteers to establish normative values for the MS-COG. A total of 150 to 200 participants in each of the 3 countries will be enrolled. The study sample will include healthy participants who are matched in age and level of education to the general MS patient population for the respective country and/or region.
Sampling Method: Non-Probability Sample
Enrollment: 467 (Actual)
Dates: Start 2014-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Selective Reminding Test (SRT) Score | Day 1
  The SRT measures verbal learning and memory. A participant is read a list of words and then asked to recall as many of the words as possible. Six learning trials are conducted, followed by a delay trial approximately 20 to 40 minutes later.
Brief Visuospatial Memory Test-Revised (BVMT-R) Score | Day 1
  The BVMT-R measures visual learning and memory. The stimulus page is presented for 10 seconds, and the participant is then asked to reproduce the designs as accurately as possible and in the same location on the page. Three learning trials are administered, followed by a delay trial approximately 20 to 40 minutes later. Immediately following the delay trial a recognition trial is administered to see whether the participant recognizes the figures that were on the display.
2- second and 3-second Paced Auditory Serial Addition Test (PASAT) Score | Day 1
  The PASAT assesses auditory information processing speed. A random series of numbers from 1 to 9, inclusive, are presented and the participant is instructed to consecutively add pairs of numbers so that each number is added to the one that immediately preceded it. In the 2- and 3- second PASAT, numbers are presented at a rate of 1 every 2 or 3 seconds, respectively.
Symbol Digit Modalities Test (SDMT) Score | Day 1
  SDMT is a screening test for cognitive impairment. Participants are given 90 seconds in which to pair specific numbers with given geometric figures using a key. Scores range from 0 to 110 (best).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (8):
- United States (4):
  - Research Site, Thornton, Colorado
  - Research site, Decatur, Georgia
  - Research Site, Latham, New York
  - Research Site, Akron, Ohio
- France (2):
  - Research site, Marseille, Bouches-du-Rhône
  - Research site, Bordeaux, Gironde
- Italy (2):
  - Research site, Milan, Milano
  - Research site, Roma, Roma